CLINICAL TRIAL: NCT03911375
Title: Stress Reduction Program Based on Mindfulness for Patients With Discopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Eduardo Anitua (Other)
Collaborators: Instituto de Investigación y Formación en Ciencias Cognitivas - Nirakara (Unknown); Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIBEA-01-EC/18/MIND
Record Dates: First submitted 2019-04-02; First posted 2019-04-11 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2021-07

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (MBSR) (Experimental): Program of 30 hours of duration divided into 9 sessions with a weekly frequency of 2.5 h and an intensive session between week 6 and 7 of the program with a duration of 7.5 hours.
  Interventions: Other: Mindfulness Based Stress Reduction (MBSR)
- Control (No Intervention): Participants assigned to the control group will follow the usual treatment, according to their diagnosis.

INTERVENTIONS:
Other: Mindfulness Based Stress Reduction (MBSR) — Psycho-educational program of stress reduction based on mindfulness. Program of 30 hours of duration divided into 9 sessions with a weekly frequency of 2.5 h and an intensive session between week 6 and 7 of the program with a duration of 7.5 hours.
  Each week the theoretical contents necessary to understand the attention development practices proposed in mindfulness-based interventions will be covered. In addition, basic concepts of the psychobiology and psychology of stress and pain are explained. The subjects will have a homework load of approximately 45 minutes per day during the duration of the intervention.
  Arms: Mindfulness Based Stress Reduction (MBSR)

SUMMARY:
This study evaluates the influence of stress on inflammation and the symptomatology of the patient with back pain. Mindfulness Based Stress Reduction (MBSR) will be used in half of participants, a validated psychopedagogical intervention for stress reduction, and the participants assigned to the control group will follow the usual treatment, according to their diagnosis.

DETAILED DESCRIPTION:
The Mindfulness based stress reduction (MBSR) is a psycho-educational program of stress reduction based on mindfulness. It consists of a program of 30 hours of duration divided into 9 sessions with a weekly frequency of 2.5 h and an intensive session between the week 6 and 7 of the program with a duration of 7.5 hours. Each week, the theoretical contents that are necessary to understand the attention development practices will be covered. In addition, basic concepts of the psychobiology and psychology of stress and pain will be explained. The subjects will have a homework load of approximately 45 minutes per day during the intervention program.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with symptomatic disc disease (Participants must provide a medical report that certifies the discopathy).
* Normal or moderate mobility
* Normal cognitive state
* Patients who have previously read and signed the informed consent.
* Patients that are capable and willing to comply with the study procedures.

Exclusion Criteria:

* Serious psychopathologies
* Suicidal thoughts.
* Deep depression
* Psychosis
* Drug addiction
* Very limited functional capacity and cognitive impairment: Patientsconfined in a bed or a chair. They need the help of a third person.
* Do not incorporate during the program any clinical, psychological or pharmacological treatments different from those ones that are normally used to controlled the pain, or any drastic changes in lifestyle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Stress change | Baseline and Six months
  Measured with the variation of cortisol in blood. These samples are obtained from a blood test that will be done to the participants before and after starting the experimental and control programs.
Variation of cytokines | Baseline and Six months
  ((TNF) -α and interleukin (IL) -1β, IL-6 and IL17), as an approximate biomarker of inflammation. Bio-chemical markers of the discopathy: Cytokines ((TNF) -α, interleukin (IL) -1β, IL-6 and IL-17). These samples are obtained from a blood test that will be done to the participants before and after starting the experimental and control programs.
Variation of the nocturnal apnea index. | Baseline and Six months
  Sleep and breathing analysis: The performance of the sleep and breathing registration tests will be carried out in the patient's home. The sleep study will be done with a validated respiratory polygraphy (BTI-APNiA®). The sleep analysis will be controlled by a sleep technician and supervised by a sleep medicine specialist. The sleep analysis will be done to the participants before and after starting the experimental and control programs.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | Baseline and Six months
  39 items scale that offers a total score of a person's level of mindfulness.
Self-Compassion Scale (SCS) | Baseline and Six months
  Evaluates the person's ability to be kind and understanding with themselves. The scale consists of 26 items scored on a 5-point likert scale.
Perceived Stress Scale (PSS) | Baseline and Six months
  Evaluates the level of perceived stress during the last month. It consists of 14 items scored on a Likert scale from 0 to 4.
DASS-21 | Baseline and Six months
  Scale designed to assess negative mood by means of three subscales: stress, anxiety and depression. The scale has 21 items scored on a Likert scale from 0 to 3.
Chronic Pain Grade Scale (CPGS; 90) | Baseline and Six months
  Scale that assesses the intensity of pain and disability caused by pain. It is a widely used measure for the evaluation of chronic musculoskeletal pain and back pain. The scale consists of 7 items scored on a Likert scale from 0 to 10.
Brief Pain Inventory (BPI) | Baseline and Six months
  It measures both the intensity of pain (sensory dimension) and the interference of pain in the patient's life (reactive dimension) in patients with chronic pain caused by osteoarthritis, back pain and cancer.
Chronic Pain Acceptance Questionnaire-Revised (CPAQ-R) | Baseline and Six months
  Instrument designed to assess the acceptance of pain. The scale consists of 20 items scored on a Likert scale from 0 to 6.
Pain Catastrophising Scale (PCS) | Baseline and Six months
  Evaluates the tendency to magnify the threat of a painful stimulus and the feeling of helplessness in the presence of pain, as well as the inability to prevent or inhibit thoughts related to pain (both before, during, and after the painful event). The scale consists of 13 items scored on a Likert scale from 0 to 4.
Brief Fatigue Inventory (BFI) | Baseline and Six months
  The objective of this scale is to assess the severity of fatigue and the impact of fatigue caused by pain in the daily functioning of people. The scale consists of 9 items scored on a scale likert type from 0 to 10.
Pain Self-Eﬃcacy Questionnaire (PSEQ) | Baseline and Six months
  Evaluates to what extent a person with pain believes they are capable of performing their daily activities regardless of their pain. The scale consists of 10 items scored on a scale likert type from 0 to 6.
Survey of Pain Attitudes - Brief (SOPA-B) | Baseline and Six months
  Evaluates the patient's attitude to seven dimensions of the experience of chronic pain: control of pain, disability associated with pain, medical cues of pain, request for help from others when in pain, medication for pain, the influence of emotions on pain and pain as an indicator of physical damage. The scale consists of 30 items scored on a Likert scale from 0 to 4.
Pain Coping Inventory (PC) | Baseline and Six months
  Instrument designed to evaluate the pain coping strategies used by patients with chronic pain. The scale consists of 34 items scored on a Likert scale from 1 to 4.
Short Form-36 Bodily Pain Scale (SF-36 BPS) | Baseline and Six months
  It is one of the eight subscales of the SF-36 questionnaire (Ware, Kosinski & Keller, 1994) designed as a generic measure of health status for population studies.
Pain and Sleep Questionnaire (PSQ) | Baseline and Six months
  Evaluates the impact of chronic pain on sleep quality. The scale consists of 8 items scored on a visual analog scale from 0 to 100.
Satisfaction with Life questionnaire (SWLS) | Baseline and Six months
  5-item brief scale designed to measure a person's overall cognitive judgments about their satisfaction with life.
WHO-5 Well Being Index | Baseline and Six months
  5 item scale designed to evaluate the subjective psychological well-being of the person.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Fundación Eduardo Anitua, Vitoria-Gasteiz, Alava
  - Instituto de Investigación y Formación en Ciencias Cognitivas - Nirakara, Madrid, Colmenarejo
  - Facultad de Psicología de la Universidad Complutense de Madrid., Madrid, Somosaguas